CLINICAL TRIAL: NCT04368169
Title: The Effects of an Aromatic Botanical Extract on Respiratory Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-4-9100
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Health

STUDY DESIGN:
Intervention Model Description: Participants are recruited through a single health practice and randomized through block randomization to one of 2 groups: botanical extract or inert control.
Who Masked: Participant, Care Provider
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatic Extract (Experimental): Participants receive the aromatic botanical extract orally every 4-6 waking hours for 3 days.
  Interventions: Dietary Supplement: Teramune Botanical Extract
- Placebo (Placebo Comparator): Participants receive the placebo matching the botanical extract orally every 4-6 waking hours for 3 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Teramune Botanical Extract — Combination blend of aromatic plant extracts in an emulsifier carrier.
  Arms: Aromatic Extract
Other: Placebo — Emulsifier carrier without active supplement ingredients.
  Arms: Placebo

SUMMARY:
This study is a randomized, double blind, placebo controlled, intervention study evaluating the effect of an aromatic botanical extract on overall respiratory health among otherwise healthy adults.

DETAILED DESCRIPTION:
After being informed about the study and providing informed consent, patients with respiratory complaints will be randomized into a double blind placebo controlled trial of the botanical extract.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-60 years
* currently experiencing respiratory symptoms
* otherwise healthy

Exclusion Criteria:

* underlying respiratory conditions
* pregnant, breastfeeding, or trying to conceive
* tobacco use in the home
* allergies to any of the ingredients

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self identify as female
Enrollment: 71 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the 44-part Wisconsin Upper Respiratory Symptom Survey (WURSS-44) at day 3. | Baseline and Day 3
  The Wisconsin Upper Respiratory Symptom Survey (WURSS-44) is a validated, self reported instrument assessing overall respiratory health. Possible scores range from 0 to 308 with lower scores indicating fewer respiratory complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie H Hawkins, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin School of Integrative Health Sciences, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No